CLINICAL TRIAL: NCT07303309
Title: Effectiveness of High-Voltage Pulsed Radiofrequency for Chronic Lumbosacral Radicular Pain: A Randomized Controlled Trial
Brief Title: Effectiveness of High-Voltage PRF for Chronic Lumbosacral Radicular Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasanuddin University (Other)
Collaborators: Faculty of Medicine, Gadjah Mada University (Unknown); Sardjito General Hospital, Yogyakarta, Indonesia (Unknown)
Responsible Party: Principal Investigator, dr. Farhan Ali Rahman, Sp. An-T.I., F.I.P., Head of Education and Training Division RSUP Dr. Sardjito/Faculty of Medicine, Public Health, and Nursing Universitas Gadjah Mada, Gadjah Mada University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 28/KEPK-RSISA/I/2025
Record Dates: First submitted 2025-12-02; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Lumbosacral Radicular Pain; Chronic Radicular Back Pain
Keywords: pain measurement; high-voltage; pulsed radiofrequency; chronic lumbosacral radicular pain; visual analogue pain scale
MeSH Terms: interventions — Pulsed Radiofrequency Treatment

STUDY DESIGN:
Intervention Model Description: Standard/Low-voltage pulsed radiofrequency (45V) was compared with high-voltage pulsed radiofrequency (60 V)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard/Low-Voltage PRF at 45 V (Active Comparator): Pulsed Radiofrequency set the voltage at 45 V.
  Interventions: Device: Pulsed Radiofrequency; Drug: Post-operative Analgesia
- High-Voltage PRF at 60 V (Experimental): Pulsed Radiofrequency set the voltage at 60 V.
  Interventions: Device: Pulsed Radiofrequency; Drug: Post-operative Analgesia

INTERVENTIONS:
Device: Pulsed Radiofrequency — A specialist performed fluoroscopy-guided monopolar Pulsed Radiofrequency (PRF) on a prone patient using a 22-gauge cannula (Cosman CC, CR type, 10 cm with a 10 mm active tip). Sensory stimulation prior to the procedure was applied at 200 Ohm, 50 Hz (threshold: 0.3 - 0.5 V), and motor stimulation at 2 Hz (threshold: 0.9 - 1.5 V). PRF was applied at a maximum temperature of 42 centigrade, with a frequency of 2 Hz, pulse width of 20 milliseconds, and a duration of 120 seconds per cycle for three cycles. An operating room nurse set the voltage at 45 V or 60 V.
  Other Names: PRF
Drug: Post-operative Analgesia — Post-procedure analgesia in both groups was provided via IV fentanyl 0.5-1 µg/kg, administered as needed for patients reporting an NRS score greater than 4. This intervention was not a primary focus of the study.
  Other Names: Rescue Analgesia; Post-operative opioid

SUMMARY:
This randomized controlled trial compared high-voltage (60 V) and low-voltage (45 V) pulsed radiofrequency (PRF) for treating chronic lumbosacral radicular pain in adult patients. The study evaluated differences in pain reduction (using the Visual Analogue Scale [VAS] and Numeric Rating Scale [NRS-11]), functional ability (using Oswestry Disability Index scores), serum Interleukin-6 levels, and overall safety. All participants received fluoroscopy-guided PRF at 42°C for three 120-second cycles and were followed for approximately 6 weeks.

DETAILED DESCRIPTION:
Consecutive patients who met the inclusion and exclusion criteria were enrolled and randomized into two groups: the intervention group (high-voltage PRF, 60 V) and the control group (low-voltage PRF, 45 V). The sample size was calculated using the Neyman-Pearson approach with a superiority hypothesis, assuming that the intervention group would achieve greater pain reduction than the control group. Accounting for an estimated 20% dropout rate, 11 participants were required per group. Patients who voluntarily withdrew from the study were excluded from analysis, whereas patients who discontinued the intervention due to adverse effects during or after the procedure were included in the analysis and reported.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 18 years old
* Numeric Rating Scale (NRS-11) ≥ 4 at screening
* Clinical diagnosis of lumbosacral radicular pain with symptom duration ≥ 12 weeks
* Insufficient response to conservative therapy, including but not limited to pharmacotherapy and/or physiotherapy

Exclusion Criteria:

* Known hypersensitivity or allergy to medication required during the study (e.g., steroid, contrast media)
* Coagulopathy, systemic infection, localized infection at needle-entry site, lumbar fracture, myelopathy, or severe organ dysfunction (e.g., renal failure, heart failure, severe respiratory diseases)
* Comorbidities that compromise valid pain assessment (e.g., post-stroke, central neuropathy, malignancy)
* Previous neurological deficits
* Pregnancy
* Refusal of participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2025-02-07 (Actual); Primary Completion 2025-04-29 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the Numeric rating scale (NRS-11) at Follow Up | Baseline (pre-intervention) through study completion, an average of 6 weeks.
  Zero is equivalent to no pain and 10 indicates the worst possible pain.
Change from Baseline in the Visual Analog Scale (VAS) at Follow Up | Baseline (pre-intervention) through study completion, an average of 6 weeks.
  The Visual Analogue Scale (VAS) is determined by measuring the distance (in millimeters) from the patient's mark on a 100mm line to the left end of the line. The left endpoint is equivalent to "no pain" and right endpoint represents the "worst imaginable pain."

SECONDARY OUTCOMES:
Change from Baseline in Oswestry's Disability Index Score at Follow Up | Baseline (pre-intervention) through study completion, an average of 6 weeks.
  The Oswestry Disability Index (ODI) was developed to evaluate the degree of disability associated with low back pain (LBP). An increase of 10% or more from the baseline ODI score is generally considered to indicate a clinically and statistically significant change in the patient's condition.
Change from Baseline in Serum Interleukin-6 at Follow Up | Baseline (pre-intervention) through study completion, an average of 6 weeks.
  A reduction or maintenance of serum interleukin-6 levels from baseline at follow-up.

OTHER OUTCOMES:
Complication and Adverse Event | From enrollment through study completion, an average of 6 weeks.
  Any complications or adverse events that occurred during the procedure or afterward up to the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Farhan A Rahman, MD, Principal Investigator — RSUP Dr. Sardjito/Faculty of Medicine, Public Health, and Nursing Universitas Gadjah Mada; Nur S Wirawan, MD, Study Director — Department of Anesthesiology, Intensive Care, and Pain Management Hasanuddin University; Muhammad R Ahmad, MD, Study Director — Department of Anesthesiology, Intensive Care, and Pain Management Hasanuddin University
Locations (1):
- RSI Sultan Agung Islamic Teaching Hospital, Semarang, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) underlying the results presented in future publication will be made available to facilitate additional research in this area. Excluding identifiers -such as names, addresses, and medical record numbers.
Supporting Information: Study Protocol, ICF
Time Frame: The IPD will be available for 5 years, starting immediately after publication.
Access Criteria: The IPD will be accessible to all individuals who have access to the Google Drive link provided in the publication.

REFERENCES:
- [Background] Deyo RA, Mirza SK. CLINICAL PRACTICE. Herniated Lumbar Intervertebral Disk. N Engl J Med. 2016 May 5;374(18):1763-72. doi: 10.1056/NEJMcp1512658. No abstract available. PMID 27144851
- [Background] Jang JN, Park S, Park JH, Song Y, Kim YU, Kim DS, Sohn JE, Park S. Output Current and Efficacy of Pulsed Radiofrequency of the Lumbar Dorsal Root Ganglion in Patients With Lumbar Radiculopathy: A Prospective, Double-blind, Randomized Pilot Study. Pain Physician. 2023 Nov;26(7):E797-E804. PMID 37976483
- [Background] Erken B, Edipoglu IS. Efficacy of High-Voltage Pulsed Radiofrequency of the Dorsal Root Ganglion for Treatment of Chronic Lumbosacral Radicular Pain: A Randomized Clinical Trial. Neuromodulation. 2024 Jan;27(1):135-140. doi: 10.1016/j.neurom.2022.10.056. Epub 2022 Dec 1. PMID 36463027